CLINICAL TRIAL: NCT05892094
Title: Comparison of the Effect of Resistance and Aerobic Training on Vasomotor Symptoms in Women in the Climacteric Period
Brief Title: Comparison of the Effect of Exercises on Vasomotor Symptoms in Middle Aged Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gizem yilmaz, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-10840098-772.02-754
Record Dates: First submitted 2023-05-17; First posted 2023-06-07 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Hot Flashes; Menopause
Keywords: Exercise; Hot flashes; Menopause; Resistance training; Aerobic exercise; Vasomotor symptoms; Quality of life; Sleep quality
MeSH Terms: conditions — Hot Flashes; Motor Activity; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Participants will participate in a 12-week full-body resistance and aerobic exercise program. It will include full body resistance exercises two days a week and aerobic exercise program three days a week. For aerobic exercise, participants will be asked to do brisk walking 3 days a week. Participants will be called regularly to monitor their participation in the aerobic exercise program. Resistance exercises sessions will be supervised by a physical therapist. Each resistance training session will include five minutes of warm-up, forty minutes of resistance training and five minutes of cool-down. Resistance exercises will consist of weight-bearing exercises performed with the participant's own body weight. Participants in the exercise group will complete the questionnaires at baseline and after 12 weeks at the end of the intervention.
  Interventions: Other: Resistance and Aerobic Training
- Control Group (No Intervention): Participants in the control group were instructed not to change their physical activity habits during 15 weeks and to avoid any other treatment for vasomotor symptoms. Participants in the control group will complete the questionnaires at baseline and after 12 weeks.

INTERVENTIONS:
Other: Resistance and Aerobic Training — For aerobic exercise, participants will do brisk walking 30 minutes in the first two weeks, 3-6. weeks will be 35 minutes, 7th and 8th weeks will be 40 minutes.The first and last 10 minutes of each walk will be said to be done at a slow pace, for the warm-up and cool-down periods. Participants will be called regularly to monitor their participation in the aerobic exercise program, and their compliance with the exercise will be checked, and they will be motivated to continue the exercises by providing the necessary information. Resistance exercises sessions will include five minutes of warm-up, forty minutes of resistance training and five minutes of cool-down. The training load will be provided by progressively increasing the repetitions. The Borg Scale will be used to adjust the exercise intensity. Rest time between sets will be 60 seconds.
  Arms: Exercise Group

SUMMARY:
Vasomotor symptoms (VMS) develop in the premenopausal period and symptoms may persist for years after menopause.Vasomotor symptoms such as hot flashes, night sweats, mood swings and sleep disturbances affect women's quality of life. There is a need for alternative treatments to reduce vasomotor symptoms due to the inadequacy of current treatments and the need for an effective treatment. Exercise is seen as a low-risk treatment to reduce vasomotor symptoms. Resistance trainig combined with aerobic training may be effective in reducing vasomotor symptoms and improving quality of life. The effects of the combination of resistance trainig 2 days a week and aerobic trainig 3 days a week on vasomotor symptoms, quality of life, sleep disturbance and depression will be investigated and compared with the control group.

DETAILED DESCRIPTION:
The climacterium, which is seen in the transition of women from the fertile period to the life stage where they lose their fertility, is seen as a natural process of aging. The World Health Organization (WHO) defines menopause as "the permanent cessation of menstruation as a result of loss of ovarian activity". The diagnosis of menopause in women is made retrospectively, usually one year after the cessation of menstrual bleeding between the ages of 45-55. The climacteric period, which consists of four phases: premenopause, menopause, perimenopause and postmenopause, covers a period of time starting around the age of 40-45 and extending to the age of 65. The premenopausal period covers the period from the onset of menstrual irregularities and the first symptoms to menopause. The first symptoms in the premenopausal period can be seen 4 years before the cessation of menstrual bleeding. Perimenopause (transition to menopause) covers premenopause, menopause and the one-year period after menopause. The postmenopausal stage, on the other hand, takes place in a long period of time from one year after menopause in women to old age. During the climacteric period, women may experience various symptoms. Vasomotor symptoms (VMS), including both daytime hot flashes and night sweats during sleep, can be experienced by middle-aged women with regular menstrual cycles, with a prevalence peaking at approximately 79% in late perimenopause. Vasomotor symptoms affects approximately 60% to 80% of women report that they feel discomfort due to vasomotor symptoms and negatively affect their quality of life. In women, these symptoms last up to 1-2 years after menopause. However, some women may experience symptoms for 10 years or longer. Vasomotor episodes are usually felt as spontaneous warmth on the chest, neck, and face of women, and this condition has often been found to be associated with sweating, anxiety, and palpitations. These symptoms can be seen as hot flashes, night sweats and facial flushing. Vasomotor symptoms interrupt women's work and daily activities and may cause sleep problems that require medical treatment. Although the cause of vasomotor symptoms is not known exactly, it is thought to develop due to hormonal changes.

Exercise is seen as a low-risk treatment to reduce vasomotor symptoms, but the evidence in the literature is inconclusive. Some observational studies have reported less VMS in physically active postmenopausal women than in sedentary women. Results from intervention studies are of low quality. The World Health Organization recommends resistance exercise twice a week for all adults. The American College of Sports Medicine (ACSM) recommends at least two days a week of resistance exercise, as well as aerobic activities three days a week. Exercise training is especially important in postmenopausal women, where decreases in muscle strength, bone mineral density and basal metabolic rate are accelerated. Previous studies, although limited, have focused on the effect of resistance training on vasomotor symptoms. In our current study, the effects of aerobic activity combined with resistance exercises on vasomotor symptoms, quality of life, sleep disturbance and depression will be investigated and compared with the control group.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 40-65
* Those who report moderate or severe vasomotor symptoms
* Those who have not received hormone replacement therapy for at least 3 months
* Maximum of 225 minutes of physical activity per week

Exclusion Criteria:

* Receiving medical treatment for menopausal symptoms in the past 2 months
* Any medical condition or physical inability to participate in exercise training
* Systolic blood pressure >160 mmHg
* Diastolic blood pressure >100 mmHg

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Physiologic female participants with vasomotor symptoms associated with menopause will be included in the study. Physiologically, the selection of the female sex is due to the fact that physiological menopause is specific to women.
Enrollment: 36 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Change in vasomotor sypmtoms | Baseline (Before intervention) and at the end of the intervention after 12 weeks
  It will be assessed with vasomotor domain of the The Menopause-specific Quality of Life (MENQOL) Questionnaire. The MENQOL assesses the impact of the menopausal symptoms and one of the four domains is vasomotor symptoms.
Change in the Menopause-specific Quality of Life (MENQOL) Questionnaire | Baseline (Before intervention) and at the end of the intervention after 12 weeks
  The MENQOL is a validated questionnaire for the assessment of menopausal women's symptoms and an effective instrument. The MENQOL is self-administered and consists of a total of 29 items in a Likert-scale format. Each item assesses the impact of one of four domains of menopausal symptoms, as experienced over the last month: vasomotor, psychosocial, physical, and sexual.
Change in the Menopause Rating Scale (MRS) | Baseline (Before intervention) and at the end of the intervention after 12 weeks
  MRS is a health-related quality of life scale (HRQoL) and was developed in response to the lack of standardized scales to measure the severity of aging-symptoms and their impact on the HRQoL. The MRS consists of a list of 11 items. Each of the eleven symptoms contained in the scale can get 0 (no complaints) or up to 4 scoring points (severe symptoms) depending on the severity of the complaints perceived by the women completing the scale.

SECONDARY OUTCOMES:
Change in the Pittsburgh Sleep Quality Index (PSQI) | Baseline (Before intervention) and at the end of the intervention after 12 weeks
  The PSQI is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Yılmaz, RA, Principal Investigator — Medipol University; Zeliha Candan Algun, PhD, Principal Investigator — Medipol University; Ahmet Fatih Durmuşoğlu, PhD, MD, Principal Investigator — Medipol University; Sebile Güler Çekiç, PhD, MD, Principal Investigator — Koç University
Locations (2):
- Turkey (Türkiye) (2):
  - Koc University Hospital, Istanbul
  - Istanbul Medipol University, Istanbul